CLINICAL TRIAL: NCT06499181
Title: Can Using Exparel Decrease the Post Operative Use of Narcotics in Maxillary Orthognathic Surgery?
Brief Title: Multimodal Orthognathic Study Comparing Use of Exparel With Standard of Care.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick Morrell, Principal Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMCSD.2017.0067
Record Dates: First submitted 2024-06-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: The control arm will be injected with 10cc of 0.5% bupivacaine with 1:50,000 epinephrine. The study arm will be injected with 133mg (10cc) of liposomal bupivacaine.
Who Masked: Participant, Care Provider
Masking Description: The control arm will be injected with 10cc of 0.5% bupivacaine with 1:50,000 epinephrine. The study arm will be injected with 133mg (10cc) of liposomal bupivacaine. Once the patient leaves the OR, the rest of the providers will be blinded to which arm the patient has been randomized. The identity will be linked to a key that will be kept in a locked box inside a keypad entry office. All future pain assessors will be blinded to the arm of the study in which the patient is attached. The patients will be taught about the surveys during the original evaluation, the consent process, and again post-operatively. An email will be sent to the patients on the following morning for the first 7 days post-operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group Exparel (Experimental): The experimental arm will be injected with 133mg (10cc) of liposomal bupivacaine (Exparel) near to the incision site one time only at the completion of the procedure.
  Interventions: Drug: Liposomal bupivacaine
- Control Group Bupivacaine (Active Comparator): The control arm will be injected with 10cc of 0.5% bupivacaine (50 mg) with 1:50,000 epinephrine near to the incision site one time only at the completion of the procedure per standard procedure.
  Interventions: Drug: Bupivacain; Drug: Epinephrin

INTERVENTIONS:
Drug: Liposomal bupivacaine — The primary objective is to examine differences in post-operative opioid consumption between the two groups.
  Other Names: Exparel
  Arms: Experimental Group Exparel
Drug: Bupivacain — Control group to receive 10cc of 0.5% bupivacaine with 1:50,000 epinephrine at the completion of the procedure per typical standard of care.
  Other Names: Marcaine, Sensorcaine
  Arms: Control Group Bupivacaine
Drug: Epinephrin — Control group to receive 10cc of 0.5% bupivacaine with 1:50,000 epinephrine at the completion of the procedure per typical standard of care.
  Other Names: Adrenalin Chloride, Epipen
  Arms: Control Group Bupivacaine

SUMMARY:
A prospective, randomized clinical trial to determine if using liposomal bupivicaine in maxillary orthognathic procedures can reduce the post-operative use of opioids as well as improving the patient's quality of life, versus traditional bupivicaine alone.

DETAILED DESCRIPTION:
A prospective randomized clinical trial to determine if using liposomal bupivicaine in maxillary orthognathic procedures can reduce the post-operative use of opioids as well as improving the patient's quality of life versus traditional bupivicaine alone. A total of 100 patients who would ordinarily undergo maxillary orthognathic procedures will be randomized into 2 groups. One group will receive 133mg of Exparel (must limit volume of product due to spaces involved and other studies in oral surgery have used 133mg) at the completion of the procedure while the control group receives 50 mg of bupivicaine at the completion of the procedure as is typical standard of care. The injections will be made in similar regions near the incision lines. No other differences will be made between the groups. Perioperative anesthesia will consist of non-opioid techniques, and patients will be monitored post-operatively during a 1 night hospital admission. Patients will complete an anonymous daily diary for 7 days. The diary will consist of information regarding pain scores, quality of life (nausea, swelling, oral function, etc) and medicines taken.

At one week post op the participant will return to the clinic where they will fill out a final questionnaire discussing the previous week's experience regarding the topics of the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Scheduled for Maxillary Orthognathic Surgery
* American Society of Anesthesiologists classification 1,2,3
* Able to provide consent, adhere to study schedule, complete study journal

Exclusion Criteria:

1 History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics or opioids.

2 Contraindication to lidocaine, epinephrine, bupivacaine, or oxycodone

3 Significant drug allergy history

4 Positive result from urine drug screen at pre-op visit

5 Currently pregnant or nursing at time of study or within 1 month of drug administration

6 Severe renal or hepatic impairment, significant cardiovascular disease; migraines, frequent headaches

7 Use of any of the following medication within 1 month of liposomal bupivacaine infiltration or if the medications are being given to control pain: Selective Serotonin Reuptake Inhibitors (SSRIs), Serotonin Nonadrenaline Reuptake Inhibitors (SNRIs), gabapentin, pregabalin, or duloxetine.

8 Current use of systemic glucocorticosteroids within 1 month of enrollment in the study.

9 No concurrent procedures with 2 weeks before or after orthognathic procedure

10 No more than 1 previous surgery for similar condition or diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Differences in post-op opioid consumption between local Exparel infiltration and bupivacaine in maxillary orthognathic procedures. | Daily up to seven days post operative procedure.
  The primary objective is to examine differences in post-operative opioid consumption between the two groups

SECONDARY OUTCOMES:
Post-operative nausea and vomiting | Daily up to seven days post operative procedure.
  Examine the number of times per day the participant experiences nausea and/or vomiting.
Post-operative sleeping quality. | Daily up to seven days post operative procedure.
  The Epworth Sleepiness Scale will be used to ascertain the quality of sleep. Eight situations are presented with the participant choosing the following responses:
  No chance of dozing = 0 Slight chance of dozing = 1 Moderate chance of dozing = 2 High chance of dozing = 3
  The higher the combined score the poorer the quality of sleep.
Post operative quality of life. | Daily up to seven days post operative procedure.
  Post operative quality of life was ascertained with the 10 point Likert scaled question, "What is your rating for your actual overall comfort?'. 1 = Very low overall comfort, 5 = Neither low or high overall comfort, 10 = Very high overall comfort.
  The higher the score means a better outcome.
Post operative oral function. | Day of surgery and at seventh day post operative procedure.
  Clinician will assess occlusion and midline symmetry on day of surgery post operative procedure and at one week post operative procedure clinic visit per standard of care with the aid of photographs using a millimeter ruler.
Post operative swelling. | Day of surgery and on post operative procedure day seven.
  Photos comparing cheek and lower jaw swelling with a millimeter ruler taken on day of surgery post operative procedure and one week post operative procedure clinic visit will be made by clinician per standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Morrell, DMD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No